CLINICAL TRIAL: NCT02555059
Title: Special Drug Use Investigation of Ciproxan® Injection in Pediatrics
Brief Title: Special Drug Use Investigation of Ciproxan Injection in Pediatrics
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18235
Record Dates: First submitted 2015-09-18; First posted 2015-09-21 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Cystitis / Pyelonephritis / Cystic Fibrosis / Anthrax
Keywords: Ciprofloxacin; Japan; Post-marketing surveillance
MeSH Terms: conditions — Cystitis; Pyelonephritis; Cystic Fibrosis; Anthrax | interventions — Ciprofloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAYQ3939: Pediatrics patients treated with Ciproxan injection in daily clinical practice.
  Interventions: Drug: Cipro (Ciprofloxacin, BAYQ3939)

INTERVENTIONS:
Drug: Cipro (Ciprofloxacin, BAYQ3939) — Treatment parameters following the physician's decision based on the summary of product characteristics.

SUMMARY:
The objective in this study is collecting post-marketing information on the safety and efficacy of Ciproxan injection under the routine clinical practice.

DETAILED DESCRIPTION:
This company-sponsored study is an one-arm, prospective, and, cohort-observational study in pediatrics (less than 15 years old) administered Ciproxan injection. All patients in the contracted institute should be enrolled into this study. Consequently 45 cases will be is planned to be enrolled in three-year period Target population is pediatrics with a diagnosis of complicated cystitis, pyelonephritis, cystic fibrosis, or anthrax infected by ciprofloxacin-active microorganisms, i.e. Bacillus anthracis, Escherichia coli, Pseudomonas aeruginosa. The treatment should be performed based on the product label in Japan. The standard observation will be performed until the last date of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female and male pediatric patients (less than 15 years old) with a diagnosis of complicated cystitis, pyelonephritis, cystic fibrosis, or anthrax infected by ciprofloxacin-active microorganisms, i.e. Bacillus anthracis, Escherichia coli, Pseudomonas aeruginosa.
* Patients for whom the decision to initiate treatment with Ciproxan injection was made as per investigator's routine treatment practice.

Exclusion Criteria:

* N/A

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Female and male pediatric patients (less than 15 years old) with a diagnosis of complicated cystitis, pyelonephritis, cystic fibrosis, or anthrax infected by ciprofloxacin-active microorganisms, i.e. Bacillus anthracis, Escherichia coli, Pseudomonas aeruginosa, are enrolled after the decision for treatment with Ciproxan injection has been made by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Number of musculoskeletal adverse events. | Up to 12 months

SECONDARY OUTCOMES:
Existence of Bacillus anthracis or Escherichia coli or Pseudomonas aeruginosa in urine(Y/N) | At week 6
Number of participants with adverse events as measure of safety and tolerability | At week 4
Efficacy | Up to 2 weeks
  Rated by physician with 3-grade scale
Number of participants with adverse events based on abnormal laboratory measurements | At week 4

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan